CLINICAL TRIAL: NCT02713373
Title: A Phase Ib/II Study of Cetuximab and Pembrolizumab in Metastatic Colorectal Cancer
Brief Title: Cetuximab and Pembrolizumab in Treating Patients With Colorectal Cancer That is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 274515; NCI-2016-00228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 274515 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2016-03-11; First posted 2016-03-18 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Colorectal Carcinoma; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Antibodies, Monoclonal; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (cetuximab and pembrolizumab) (Experimental): Patients receive cetuximab IV over 120 minutes on day 1 (days 1, 7, and 14 of course 1 only) and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity. Patients may continue pembrolizumab treatment for up to 1 year if they experience disease progression.
  Interventions: Biological: Cetuximab; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-Epidermal Growth Factor Receptor (EGFR) Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/II trial studies the side effects and best dose of cetuximab when given together with pembrolizumab in treating patients with colorectal cancer that has spread from the primary site (place where it started) to other places in the body (metastatic) or that cannot be removed by surgery. Monoclonal antibodies, such as cetixumab and pembrolizumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the objective response rate of patients with metastatic colorectal cancer treated with pembrolizumab and cetuximab.

II. To estimate the 6-month progression free survival (PFS) rate of patients with metastatic colorectal cancer treated with pembrolizumab and cetuximab.

III. To examine the adverse event profile of combining pembrolizumab and cetuximab.

SECONDARY OBJECTIVES:

I. To examine the PFS of patients with metastatic colorectal cancer treated with pembrolizumab and cetuximab.

II. To determine the objective response rate by immune-related response criteria (irRC) of patients with metastatic colorectal cancer.

III. To examine the overall survival of patients with metastatic colorectal cancer treated with pembrolizumab and cetuximab.

EXPLORATORY OBJECTIVES:

I. Identify tumor and peripheral blood biomarkers of response and/or resistance to the study treatment.

OUTLINE:

Patients receive cetuximab intravenously (IV) over 120 minutes on day 1, 8, and 15 (as monotherapy for cycle 1 only) and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity. Patients may continue pembrolizumab treatment for up to 1 year if they experience disease progression.

After completion of the study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a pathologically confirmed diagnosis of colorectal cancer, which is metastatic or otherwise unresectable
* Have received at least 1 prior systemic therapy in the metastatic or unresectable disease setting; patients who have recurred within six months of adjuvant chemotherapy are not required to have received an additional line of chemotherapy
* Retrovirus-associated deoxyribonucleic acid (DNA) sequence (RAS) wild-type; v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) testing must be completed, with full KRAS and neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS) testing strongly advised; the presence of known mutations in KRAS or NRAS is exclusionary; primary tumor or metastatic tumor may be tested; (note: in the case of multiple genomic evaluations with conflicting results - e.g. KRAS mutant in one sample, but wild-type in another - the patient may be included as RAS wild-type, if clinically justified, after review with the principal investigator [PI])
* Appropriate for anti-EGFR therapy: Naive to anti-EGFR therapy (cetuximab or panitumumab) or a candidate for rechallenge by virtue of the following:

  1. the investigator deems anti-EGFR retreatment with cetuximab to be a reasonable standard of care option AND
  2. outcome of prior anti-EGFR therapy was not rapid progression (i.e. <= 3 months on therapy) AND
  3. prior anti-EGFR therapy was administered > 6 months prior to the start of protocol therapy
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion; newly-obtained is defined as a specimen obtained up to 30 days prior to initiation of treatment on day 1
* Hemoglobin >= 8 g/dL (performed within 14 days of treatment initiation)
* Absolute neutrophil count >= 1000/mm3 (performed within 14 days of treatment initiation)
* Platelet count >= 100,000/mm3 (performed within 14 days of treatment initiation)
* Serum creatinine =< 2 upper limit of normal (ULN) or, >= 15 mL/min for participants with creatinine levels > 2 ULN (performed within 14 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 ULN or, =< 5 ULN for participants with liver metastases (performed within 14 days of treatment initiation)
* Female participants of childbearing potential are to have a negative serum pregnancy test
* Female participants of child-bearing potential must agree to use an acceptable method of birth control, be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants who have had chemotherapy, targeted therapies, radiotherapy, or used an investigational device within 2 weeks prior to the first dose of treatment or those who have not recovered from adverse events (i.e., =< grade 1 or at baseline) due to agents administered more than 2 weeks earlier; note: participants with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Prior severe infusion reaction to cetuximab
* Has a known additional malignancy that requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Uncontrolled clinically significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness, substance abuse disorders or social situations that would limit compliance with study requirements
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV or HIV 1/2 antibodies); testing not required
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected); testing not required
* Has received a live vaccine within 30 days of planned start of study therapy (note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and shingles are not allowed)
* Received an investigational agent within 30 days prior to starting study treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five patients were enrolled in our study; one patient was not treated secondary to clinical progression during the screening period
Period: Overall Study
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Examine the Adverse Event Profile
Description: The frequency of toxicities will be tabulated by maximum grade by preferred term within a patient across all cycles.
Time Frame: up to 24 months
Measure: Number; unit: participants
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
participants
  Dry skin | 21
  acneiform dermatitis | 20
  fatigue | 17
  hypomagnesemia | 16
  rash | 16
  diarrhea | 12
  pruritus | 12
  anorexia | 10

2. Primary Outcome: Progression Free Survival (PFS), Evaluated According to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), At least a 20% increase in the sum of diameters of target lesions, taking as references the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: percentage of PFS at 6 months
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
percentage of PFS at 6 months | 31 [20 to 43]

3. Primary Outcome: Number of Participants With a Response, Evaluated According to RECIST 1.1
Description: Number of Participants with a Response, Evaluated According to RECIST 1.1 will be tabulated and will be compared to the null values using exact tests.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
Participants | 1

4. Secondary Outcome: Objective Tumor Response Using Immune-related RECIST
Description: tumor response using immune-related RECIST (irRECIST) will be tabulated, summarized and reported.
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
Participants
  PD Progressive Disease | 11
  PR Partial Response/Remission | 1
  SD Stable Disease | 27
  TE Too Early | 1
  NE Not Evaluable | 3
  OT Other | 1

5. Secondary Outcome: Overall Survival (OS)
Description: Distributions of OS will be estimated using the Kaplan-Meier method.
Time Frame: Up to death, withdrawal of consent, or the end of the study, whichever occurs first, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
months | 14.5 [11.6 to 19.6]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Distributions of PFS will be estimated using the Kaplan-Meier method. Median PFS is reported.
Time Frame: Up to15 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
Number analyzed (Participants) | 44
Months | 4.1 [3.9 to 6.0]

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | Arm I (Cetuximab and Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 32/44
Serious Adverse Events (participants affected / at risk) | 9/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cetuximab and Pembrolizumab) (N=44)
Constipation (Gastrointestinal disorders) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urosepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cetuximab and Pembrolizumab) (N=44)
Anaemia (Blood and lymphatic system disorders) | 7 (26)
Lymphopenia (Blood and lymphatic system disorders) | 2 (4)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Eye disorder (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Visual impairment (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 14 (22)
Diarrhoea (Gastrointestinal disorders) | 15 (26)
Dry mouth (Gastrointestinal disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (20)
Oral pain (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 9 (14)
Catheter site related reaction (General disorders) | 1 (1)
Chills (General disorders) | 6 (6)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 18 (31)
Influenza like illness (General disorders) | 1 (1)
Infusion site reaction (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 5 (5)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 7 (8)
Tenderness (General disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (10)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (14)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Blood alkaline phosphatase (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (6)
Blood bilirubin increased (Investigations) | 2 (3)
Blood creatinine increased (Investigations) | 3 (23)
Blood magnesium decreased (Investigations) | 2 (2)
Carbon dioxide decreased (Investigations) | 1 (1)
International normalised ratio (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (3)
Lymphocyte count decreased (Investigations) | 4 (11)
Lymphocyte count increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Transaminases increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Weight increased (Investigations) | 1 (3)
White blood cell count decreased (Investigations) | 1 (4)
Decreased appetite (Metabolism and nutrition disorders) | 10 (17)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 (54)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5)
Drooling (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Sciatica (Nervous system disorders) | 1 (2)
Taste disorder (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (12)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 20 (32)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (26)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 3 (3)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 7 (7)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 (3)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (14)
Rash (Skin and subcutaneous tissue disorders) | 16 (24)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT02713373/Prot_SAP_000.pdf